CLINICAL TRIAL: NCT02870179
Title: Oxitone Sp02 Hypoxia Test Versus Reference Pulse Oximetry
Status: Completed | Type: Observational
Sponsor: Oxitone Medical Ltd. (Industry)
Collaborators: Clinimark, LLC (Other)
Responsible Party: Principal Investigator, Leon Eisen, PhD, Leon Eisen, CEO, Oxitone Medical Ltd.
Other Study IDs: PR 2016-191
Record Dates: First submitted 2016-08-10; First posted 2016-08-17 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Hypoxia
Keywords: Pulse Oximetry; Temperature; Respiratory Rate; Respiratory Gases; This study determines the measurement accuracy of the physiological parameters
MeSH Terms: conditions — Hypoxia | interventions — Blood Pressure; Respiratory Rate; Body Temperature

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy volunteer: Smoker or non-smoker
  Interventions: Device: Pulse Oximeter

INTERVENTIONS:
Device: Pulse Oximeter — Measurement of physiological parameters
  Other Names: Blood Pressure; Respiratory Rate; Respiratory Gassess; Temperature

SUMMARY:
The purpose of this study is to conduct a SpO2 hypoxia evaluation of the Oxitone Medical Oxitone 1000 pulse oximeter. The Oxitone 1000 pulse oximeter will be evaluated during non-motion conditions over the range of 70-100% SpO2 in comparison to a Reference Pulse Oximeter.

The study is observational in nature which quantifies device performance and accuracy in compassion to a Reference Pulse Oximeter.

DETAILED DESCRIPTION:
The purpose of this study is to conduct a SpO2 hypoxia evaluation of the Oxitone Medical Oxitone 1000 pulse oximeter. The Oxitone 1000 pulse oximeter will be evaluated during non-motion conditions over the range of 70-100% SpO2 in comparison to a Reference Pulse Oximeter. The end goal is to show the SpO2 accuracy performance of the Oxitone 1000 and if needed, use the data to make improvements prior to an arterial blood hypoxia study.

A Clinimark 3900 Reference Pulse Oximeter or Nellcor N-600x will be used for the SpO2 calibration. There are no risks or adverse device effects to be assessed. There are no contraindications for use in the proposed study / study population

The Control Pulse Oximeter, GE Healthcare (Datex-Ohmeda) 3900, an FDA cleared device, is used to monitor the oxygen saturation levels real time throughout the study for subject safety and to target stable plateaus. This device is used to assess the stability of the data.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals between the age of 18-50

Exclusion Criteria:

* Clotting disorders, diabetes, currently taking psychotropic medications

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Residents of the Denver metropolitan area
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Collect SpO2 data for accuracy statistical analysis by 12 subjects | 2 months
  Data is collected in a digital form for 4-6 SpO2 stable plateaus in a specified range from 100% to 70%.
Accuracy data analysis | 2 months
  Bland-Altman graphical plots. An Accuracy Root Mean Square (ARMS) calculation is used as a means to define the SpO2 accuracy. Data analysis will follow ISO80601-2-61, Annex EE and the FDA Guidance Document for Pulse Oximeters (Martch 4, 2013).

SECONDARY OUTCOMES:
Error plots | 2 months
  SpO2 versus (SpO2-Ref SpO2) will be generated with linear regression fit, mean, and upper 95% and lower 95% limits of agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Leon Eisen, PhD, Principal Investigator — Oxitone Medical Ltd.
Locations (1):
- Clinimark Laboratories, Louisville, Colorado, United States